### **Addendum Study**

# Telehealth Study Assessing Filter Ventilation on Smoking Behavior and Biomarkers Consent Form for Inhalation Study

You are invited to participate in an addendum research project conducted by Dorothy Hatsukami, Ph.D. at the University of Minnesota's Masonic Cancer Center and Peter Shields, MD at The Ohio State University.

# Why am I being asked to take part in this research study?

We are asking you to take part in this research study because you are participating in the "Telehealth Study Assessing Filter Ventilation on Smoking Behavior and Biomarkers"

# Why is this research being done?

We are studying the effects of filter ventilation on how you inhale your cigarette.

## How long will the research last?

You will have the inhalation measures done twice during the study, once on the day you start your randomized study cigarettes and once when you finish smoking the study cigarettes.

#### **Procedures**

If you agree to participate in the addendum Inhalation Study, we will conduct a procedure that measures how you inhale and exhale your cigarette while smoking. For this inhalation test, you will have two bands, one placed around your chest and one around your abdomen. These bands are connected to a computer program that will measure your breaths while smoking. This procedure will take less than 30 minutes at the two visits.

### What happens if I do not want to be in this research?

This is a research study and you can choose whether or not you want to participate. You can stop participating in the Inhalation Study and still continue with the main study.

#### **Risks and Benefits**

You will receive no direct benefit form your participation in this study. There are no additional risks in participating in this study.

# Will I be compensated for my participation?

You will receive an additional \$25 on your Clincard for each inhalation session.

<u>Please review your Consent Form for the main study for contact and other applicable</u> information.

IRB# 00012328

Addendum Version date: 05AUG2021

| You are making a decision whether or not to participate. Your signature indicates that you have read the information provided above and you have decided to participate. You may withdraw from the study at any time without prejudice after signing this form You will be provided with a copy of this form to keep. Statement of consent Your signature below documents your permission to take part in this research. You will be provided a copy of this signed document. | | | |
|---|---|---|---|
| | | Signature of Participant | Date |
| | | Printed Name of Participant | |
| Signature of Staff Obtaining Consent | <br>Date | | |

Addendum Version date: 05AUG2021

Printed Name of Staff Obtaining Consent